CLINICAL TRIAL: NCT06412601
Title: Happy Bob App: A Preliminary Evaluation of Its Use in Youth With Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jacob Redel, Physician, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002907
Record Dates: First submitted 2024-04-18; First posted 2024-05-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RPM (remote patient monitoring) (Experimental)
  Interventions: Behavioral: RPM; Behavioral: app
- Non-RPM (Active Comparator)
  Interventions: Behavioral: app

INTERVENTIONS:
Behavioral: RPM — remote patient monitoring by clinic staff
  Arms: RPM (remote patient monitoring)
Behavioral: app — use of Happy Bob phone app

SUMMARY:
The goal of this clinical trial is to evaluate the impact of peer support via the Happy Bob phone app in youth with Type 1 Diabetes.

The main questions it aims to answer are: What is the usability and acceptability of the app? What is the app's efficacy on measures such as treatment adherence and social support? And how are these effects impacted by remote patient monitoring by clinic staff?

Participants will use the Happy Bob app for 6 months and will complete a series of surveys at the start, middle, and end of their use of the app. Some participants will participate in 2 remote patient monitoring sessions when beginning their use of the app.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Type 1 Diabetes, Use Dexcom and Smart Phone

Exclusion Criteria:

Non-English Speaking

Ages: 13 Years to 215 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Happy Bob App User Metrics | 6 months
  time spent in Happy Bob,
Type 1 Diabetes and Life (T1DAL) Measure | 0,3,6 months
  quality of life scale
Positive and Negative Affect Schedule (PANAS) | 0,3,6 months
  mood scale
Diabetes Treatment Satisfaction Questionnaire | 0,3,6 months
  intervention satisfaction
Social Support Questionnaire for Children (SSQC) | 0,3,6 months
  social quality of life
Health Information Technology Usability Evaluation Scale (Health-ITUES) | 0,3,6 months
  usability scale

SECONDARY OUTCOMES:
Self Efficacy for Diabetes (SED) Scale | 0,3,6 months
  efficacy scale
Diabetes Treatment Outcomes | 6 months
  TIR,

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No